CLINICAL TRIAL: NCT02618889
Title: OnabotulinumtoxinA in the Management of Psychogenic Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alberto Espay, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-4496
Record Dates: First submitted 2015-10-21; First posted 2015-12-02 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Torticollis, Dystonia
MeSH Terms: conditions — Torticollis; Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT plus botox (Active Comparator): Participants will be randomized to receive BoNT (onabotulinumtoxinA). Patients will undergo study assessments four weeks later. We will inject a total of 250 units of onabotulinumtoxinA, as the average optimal dose in cervical dystonia,11 using a 100:1 dilution with normal saline. The target muscles will be the ones deemed most active in the cervical region or in any of the affected limbs. If several limbs are affected, only up to two will be targeted in similar fashion, with a total dose not to exceed 400 units altogether (250 +150 units, if involvement is asymmetric or unilateral [leg and arm, respectively]; 200 + 200 units, if involvement is symmetric).
  Interventions: Behavioral: CBT
- CBT plus placebo (Placebo Comparator): Participants will be randomized to receive normal saline (placebo). We will inject a total of 250 units of normal saline, as this is the average optimal dose of onabotulinumtoxinA in cervical dystonia. The target muscles will be the ones deemed most active in the cervical region or in any of the affected limbs. If several limbs are affected, only up to two will be targeted in similar fashion, with a total dose not to exceed 400 units altogether (250 +150 units, if involvement is asymmetric or unilateral [leg and arm, respectively]; 200 + 200 units, if involvement is symmetric).
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — All participating subjects will start a 12-week CBT treatment program. These consist of weekly 1-hour CBT sessions led by a cognitive therapist. Assessments will be repeated at week 16. All PsyD subjects will undergo a 15-minute, structured diagnostic interview (Mini International Neuropsychiatric Interview (MINI)) developed to screen for axis I DSM-IV and ICD-10 psychiatric disorders. We will also use two clinician-rated instruments to assess comorbid psychopathology in PsyD patients, the 17-item Hamilton Depression Rating Scale (HAM-D), to evaluate for depressed mood, vegetative and cognitive symptoms of depression; and the 14-item Hamilton Anxiety Rating Scale (HAM-A) to evaluate psychic and somatic anxiety. These scales will be administered as part of a structured interview.

SUMMARY:
The purpose of this research study is to evaluate if patients with psychogenic dystonia treated with onabotulinumtoxinA (BOTOX) injections will demonstrate lower severity and disability at one month and at three months than those having received placebo injections

DETAILED DESCRIPTION:
Specific Aim 1: To investigate the effect of BoNT on PsyD severity and disability.

We will measure the changes in severity, duration, and incapacitation scores of the Rating Scale for Psychogenic Movement Disorders (RSPMD)10 in adult patients with clinically definite PsyD one month after intramuscular injections with onabotulinumtoxinA in selected muscles of the affected limb(s).

H1: PsyD patients treated with onabotulinumtoxinA injections will demonstrate lower severity and disability at one month than those having received placebo injections.

Specific Aim 2: To investigate the effect of CBT on PsyD severity and disability with and without BoNT pretreatment.

We will examine the extent to which any changes in severity and disability of PsyD, as measured by the RSPMD, after 12 weekly CBT sessions, can be influenced by pre-CBT injections with onabotulinumtoxinA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet standard criteria for clinically definite PsyD;17
* PsyD severity and disability score ≥ 10 as measured by the RSPMD (Appendix 1);10
* Dystonic posturing must have been present without remission for a period longer than 1 year.
* Between the ages of 18 and 75, inclusive

Exclusion Criteria:

* Prior treatment with any BoNT
* Presence of clinically unstable medical condition other than the condition under evaluation
* Concurrent participation in another investigational drug or device study within 30 days prior to study enrollment.
* We will also exclude subjects with medical disorders deemed at increased risk when exposed to BoNT, including myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or other neuromuscular disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Rating Scale for Psychogenic Movement Disorders (RSPMD) | 4 months
  Primary outcome measures will be the combined severity, duration factor, and incapacitation scores (investigator-rated) of the Rating Scale for Psychogenic Movement Disorders (RSPMD, 0-12 per each limb and head [maximum for all five regions: 60]) (see Appendix 1).

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) of change | 4 months
  7-point Likert scale ("very much improved," to "very much worse")
Hamilton Depression Rating Scale (HAM-D) | 4 months
  neuropsychiatric measures of depression.
Hamilton Anxiety Rating Scale (HAM-A) | 4 months
  neuropsychiatric measures of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Espay, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Alberto Espay, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No